CLINICAL TRIAL: NCT04145635
Title: An Evaluation of the Safety and Performance of the Aortix System for Intra-Aortic Mechanical Circulatory Support in Patients With Cardiorenal Syndrome
Brief Title: The Aortix CRS Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Procyrion (Industry)
Collaborators: Procyrion Australia Pty Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PVP017
Record Dates: First submitted 2019-10-25; First posted 2019-10-30 (Actual); Results first posted 2024-04-17 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Heart Failure; With Decompensation; Cardiorenal Syndrome; Cardio-Renal Syndrome; Heart Failure; Heart Failure，Congestive; Heart Failure, Systolic; Heart Failure, Diastolic
Keywords: mechanical circulatory support, percutaneous
MeSH Terms: conditions — Heart Failure; Cardio-Renal Syndrome; Heart Failure, Systolic; Heart Failure, Diastolic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Aortix Device (Experimental): Aortix Pump, Aortix Delivery System, Introducer Set, Aortix Control System, Aortix Retrieval System
  Interventions: Device: Aortix System

INTERVENTIONS:
Device: Aortix System — Aortix is a circulatory support device for chronic heart failure patients on medical management who have been hospitalized for acute decompensated heart failure (ADHF) with worsening renal function.

SUMMARY:
The Aortix CRS Pilot Study: An Evaluation of the Safety and Performance of the Aortix System for Intra-Aortic Mechanical Circulatory Support in Patients with Cardiorenal Syndrome

DETAILED DESCRIPTION:
The study is a prospective, multi-center, non-randomized feasibility study to evaluate the safety and performance of the Aortix System in patients hospitalized with acute decompensated heart failure (ADHF) and worsening renal function refractory to medical management with persistent congestion. The Aortix system consists of the Aortix Delivery System, Introducer Set, the Aortix Pump, the Aortix Control System, and the Aortix Retrieval System.

ELIGIBILITY:
Inclusion Criteria:

1) Admitted to the hospital with a primary diagnosis of acute decompensated heart failure, either heart failure with reduced or preserved ejection fraction (HFrEF, HFpEF or HFmEF);

2) Worsening renal function (serum creatinine increase by ≥0.3 mg/dl [≥27 μmol/L]) despite 48 hours of intravenous diuretic therapy Increase can be compared to a baseline value taken within 90 days of hospitalization or during hospitalization;

3) Objective measure of congestion (Elevated PCWP [≥20 mmHg] OR Elevated CVP [≥12 mmHg]) obtained via catheter measurement;

4) Persistent clinical signs and/or symptoms of congestion despite diuretic therapy (one or more of the following):

1. dyspnea at rest or with minimal exertion,
2. paroxysmal nocturnal dyspnea,
3. orthopnea,
4. lower extremity edema (≥2+),
5. elevated jugular venous pressure,
6. pulmonary rales,
7. enlarged liver or ascites,
8. pulmonary vascular congestion on chest x-ray;

   5) Age >21 years.

   -

   Exclusion Criteria:

   1) Treatment with high dose IV inotropes within the last 48 hours. High dose is defined as > 1 unit of inotrope (excluding digoxin) as follows: 5 µg/kg/min dopamine = 1 unit, 5 µg/kg/min dobutamine= 1 unit, 0.375 µg/kg/min milrinone = 1 unit, (for example, dopamine 2.5 µg/kg/min + dobutamine 2.5 µg/kg/min = 1 unit; dobutamine 2.5 µg/kg/min + milrinone 0.1875 µg/kg/min = 1 unit);

   2) Treatment with vasopressors to maintain blood pressure as per exclusion number 3;

   3) Active and ongoing hypotension defined as a systolic blood pressure < 90 mmHg lasting more than 30 minutes or a mean arterial pressure (MAP) < 60 mmHg lasting more than 30 minutes;

   4) Acute Kidney Failure defined as increase in serum creatinine to ≥4.0 mg/dL (≥353.6 μmol/L) within the last 48 hours;

   5) Exposure to intravenous contrast, aminoglycosides or high dose NSAIDS in the 48 hours before enrollment;

   6) Known or suspected contrast induced nephropathy;

   7) Prior kidney transplant, isolated single kidney, stage V Chronic Kidney Disease (eGFR ≤15) at admission OR use of dialysis, continuous renal replacement therapy (CRRT) or aquapheresis (ultrafiltration) in last 90 days;

   8) Urologic intervention (except indwelling urinary (Foley) catheter)) within the last 7 days;

   9) Known cirrhosis or shock liver;

   10) Presence of an active infection;

   11) Prior heart transplant in the last 2 years, heart failure due to rejection of a previous heart transplant, planned heart transplantation before the 30-day follow-up visit;

   12) Current or previous support with a durable LVAD at any time or use of an intra-aortic balloon pump, extracorporeal membrane oxygenation (ECMO), or percutaneous ventricular assist devices (e.g. Impella or TandemHeart) currently or within the last 30 days;

   13) Patient has known hypo- or hyper coaguable state such as disseminated intravascular coagulation or heparin induced thrombocytopenia (HIT);

   14) Known cardiac amyloidosis;

   15) Acute myocardial infarction Type 1 within 30 days of enrollment, or planned coronary revascularization;

   16) Stroke within 30 days of enrollment;

   17) Severe Bleeding Risk (any of the following):

a) Previous intracranial bleed unless there is documentation in the medical record (from a physician that is not part of the study) that the patient can safely use anticoagulation for 7 days, b) GI bleeding within 6 months requiring hospitalization and/or transfusion, c) Recent major surgery within 6 months if the surgical wound is judged to be associated with an increased risk of bleeding, d) Endovascular procedure with ilio-femoral access > 6 FR within 30 days, e) Platelet count <75,000 cells/mm3, f) Uncorrectable bleeding diathesis or coagulopathy (e.g. INR ≥2 not due to anticoagulation therapy);

18) Current endovascular stent graft in the descending aorta or any femoro-iliac vessels;

19) Contraindicated Anatomy:

1. Descending aortic anatomy that would prevent safe placement of the device [<18mm or >31mm aorta diameter at deployment location (measured between the superior aspect of the T10 vertebra and superior aspect of the L1 vertebra)],
2. Abnormalities of the aorta or iliac arteries that would prevent safe device placement, including aneurysms, significant tortuosity, or calcifications,
3. Ilio-femoral diameter or peripheral vascular anatomy that would preclude safe placement of a 21F (outer diameter) introducer sheath including severe obstructive calcification or severe tortuosity,
4. Known connective tissue disorder (e.g. Marfan Syndrome) or other aortopathy at risk of vascular injury;

   20) Known hypersensitivity or contraindication to study or procedure medications (e.g.

   anticoagulation therapy) or device materials (e.g. history of severe reaction to nickel or nitinol);

   21) Positive pregnancy test if of childbearing potential;

   22) Participation in any other clinical investigation that is likely to confound study results or affect the study;

   23) Unable or unwilling to undergo screening (imaging, PA Catheter placement), device implant and retrieval procedures.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2021-02-05 (Actual); Primary Completion 2022-10-07 (Actual); Study Completion 2023-03-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (19):
- United States (14):
  - University of Southern California, Los Angeles, California
  - University of California, San Francisco, San Francisco, California
  - University of Colorado, Denver, Colorado
  - University of Florida, Gainesville, Florida
  - University of South Florida, Tampa, Florida
  - Cleveland Clinic Florida, Weston, Florida
  - University of Chicago, Chicago, Illinois
  - University of Michigan, Ann Arbor, Michigan
  - Henry Ford Health System, Detroit, Michigan
  - Columbia University/New York Presbyterian, New York, New York
  - Christ Hospital, Cincinnati, Ohio
  - Houston Methodist, Houston, Texas
  - Inova Health Care Services, Falls Church, Virginia
  - Sentara Hospital, Norfolk, Virginia
- Australia (5):
  - St. Vincent's Hospital, Sydney, New South Wales
  - Prince Charles Hospital, Brisbane, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - The Alfred Hospital, Melbourne, Victoria
  - Western Health, Footscray Hospital, Melbourne, Victoria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cowger JA, Basir MB, Baran DA, Hayward CS, Rangaswami J, Walton A, Tita C, Minear S, Hakemi E, Klein L, Cheng R, Wu R, Mohanty BD, Heuring JJ, Neely E, Shah P; Aortix CRS Pilot Study Investigators. Safety and Performance of the Aortix Device in Acute Decompensated Heart Failure and Cardiorenal Syndrome. JACC Heart Fail. 2023 Nov;11(11):1565-1575. doi: 10.1016/j.jchf.2023.06.018. Epub 2023 Oct 4. PMID 37804307

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Aortix Device
Started | 21
Completed | 18
Not Completed | 3

BASELINE CHARACTERISTICS:
Arm/Group | Aortix Device
Number analyzed (Participants) | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 9
  >=65 years | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.3 (7.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 10
Race/Ethnicity, Customized [Number; unit: participants]
  White | 15
  Black/African | 3
Region of Enrollment [Number; unit: participants]
  United States | 17
  Australia | 1
Baseline Ejection Fraction (%) [Median (Inter-Quartile Range); unit: %] | 22.5 [10 to 53.5]

OUTCOME MEASURES:

1. Primary Outcome: Serious Adverse Events
Description: Rate of Occurrence of Serious Adverse Events (rate will be calculated and reported)
Time Frame: 30 days
Measure: Number; unit: Events
Arm/Group | Aortix Device
Number analyzed (Participants) | 18
Events | 18

2. Primary Outcome: Serious Procedure Related Adverse Events
Description: Rate of Occurrence of Serious Procedure Related Adverse Events (rate will be calculated and reported)
Time Frame: 30 days
Measure: Number; unit: Events
Arm/Group | Aortix Device
Number analyzed (Participants) | 18
Events | 7

3. Primary Outcome: Device Performance
Description: Deployment and retrieval procedures success rates (rates will be calculated and reported).
Time Frame: 7 days
Measure: Number; unit: percentage of subjects
Arm/Group | Aortix Device
Number analyzed (Participants) | 18
percentage of subjects
  Implant Success Rate | 100
  Retrieval Success Rate | 100

4. Primary Outcome: Device Performance
Description: Rate of occurrence of ADS, ARS and pump device-related adverse events (includes device malfunctions) (rate will be calculated and reported)
Time Frame: 30 days
Measure: Number; unit: event
Arm/Group | Aortix Device
Number analyzed (Participants) | 18
event | 1

5. Primary Outcome: Effectiveness
Description: Clinically significant decongestion as measured by the PA catheter. % of patients with a decrease in either CVP or PCWP of > 20%.
Time Frame: 7 days
Measure: Number; unit: % of patients with specified decrease
Arm/Group | Aortix Device
Number analyzed (Participants) | 18
% of patients with specified decrease | 89

6. Primary Outcome: Urine Output
Description: Change in Urine Output Assessed as the hourly rate of urine output before pump placed vs hourly rate of urine output over the Aortix therapy period (until congestion target met or therapy deemed ineffective)
Time Frame: 7 day period starting from implant
Population: Patients Receiving Aortix Device
Measure: Median (Full Range); unit: mL/hr of Urine Output
Arm/Group | Aortix Device
Number analyzed (Participants) | 18
mL/hr of Urine Output
  Baseline Hourly Urine Output | 113.7 [76.0 to 167.1]
  Peak Urine Output During Treatment | 236 [177.4 to 293.8]

7. Primary Outcome: NT-pro-BNP (Brain Natriuretic Peptide)
Description: Change in NT-pro-BNP (pre-implant vs when congestion target is met or therapy deemed ineffective)
Time Frame: 7 days
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | Aortix Device
Number analyzed (Participants) | 17
pg/mL | -1,763 [-3,613 to 180]

ADVERSE EVENTS:
Time Frame: 2 years; timeframe is from enrollment to 30-day visit.
Arm/Group | Aortix Device
All-Cause Mortality (participants affected / at risk) | 2/21
Serious Adverse Events (participants affected / at risk) | 11/21
Other Adverse Events (participants affected / at risk) | 11/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aortix Device (N=21)
Arrest, Cardiac (Cardiac disorders) | 1 (1)
Bleeding/Femoral Access (Vascular disorders) | 4 (4)
Pulmonary Embolism (Vascular disorders) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 1 (1)
Thrombotic Vascular Complication (Vascular disorders) | 2 (2)
Bleeding, GI Bleed (Vascular disorders) | 1 (1)
Vascular Injury (NonAorta) (Vascular disorders) | 2 (2)
Device Migration/Dislodgement (Product Issues) | 1 (1)
Hemolysis (Vascular disorders) | 1 (1)
Hepatic Dysfunction (Renal and urinary disorders) | 1 (1)
Hypotension (Cardiac disorders) | 1 (1)
Renal Injury, AKIN Stage 2 (Renal and urinary disorders) | 1 (1)
Worsening Heart Failure (Cardiac disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aortix Device (N=21)
Bleeding Event (Vascular disorders) | 2 (2)
GI Miscellaneous (Gastrointestinal disorders) | 2 (2)
Hemolysis (Blood and lymphatic system disorders) | 7 (7)

LIMITATIONS AND CAVEATS:
Larger samples and a study powered to allow comparison with SOC is needed to confirm decongestion and renal benefits from IAEP and to identify a HF pt group that would benefit the most. An 18F sheath is required for device deployment, pts require systemic anticoagulation, and ICU monitoring was required. The implant procedure should be validated with various operators; the efficacy, performance, and safety of IAEP should be studied in a RCT; and consider extra costs of therapy vs pt outcomes.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-07-24): https://cdn.clinicaltrials.gov/large-docs/35/NCT04145635/Prot_000.pdf
  • Statistical Analysis Plan (2022-03-23): https://cdn.clinicaltrials.gov/large-docs/35/NCT04145635/SAP_003.pdf